CLINICAL TRIAL: NCT03938844
Title: Which Anti-İncontinence Surgery Option is Better in Patients With Total Laparoscopic Hysterectomy? BURCH Colposuspension or Transobturatuar Tape (TOT)
Brief Title: BURCH Colposuspension or Transobturatuar Tape (TOT)
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.01.07
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Incontinence
Keywords: hysterectomy; anti-incontinence surgery; Burch; Tot; stress incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TLH with BURCH Colposuspension: the patients who underwent simultaneous burch copying with TLH was evaluated. In addition to demographic data and preoperative examination findings, operative times, postoperative hemogram values, postvoiding residual amounts and complications were examined. In addition, FSI test results of women with sexual activity were compared with ICIQ-UI and UDI-6 interrogations related to urinary incontinence.
  Interventions: Procedure: BURCH Colposuspension
- TLH with Transobturatuar Tape (TOT): In cases of simultaneous toting with TLH; In addition to demographic data and preoperative examination findings, operative times, postoperative hemogram values, postvoiding residual amounts and complications were examined. In addition, FSI test results of women with sexual activity were compared with ICIQ-UI and UDI-6 interrogations related to urinary incontinence.
  Interventions: Procedure: TOT

INTERVENTIONS:
Procedure: BURCH Colposuspension — stress urinary incontinence surgery ( burch or tot)
  Groups: TLH with BURCH Colposuspension
Procedure: TOT
  Groups: TLH with Transobturatuar Tape (TOT)

SUMMARY:
Stress urinary incontinence surgery combined with hysterectomy can often be applied to patients in the same session. The aim of this study was to determine which urinary incontinence surgery would be a better option for patients who would have hysterectomy.

The aim of this study was to retrospectively review the data of 69 patients between the ages of 2014 and 2017 who underwent total laparoscopic hysterectomy and anti-incontinence surgery (TOT and Burch) for benign indications (uterine pathology) and stress urinary incontinence (SUI). In addition to demographic data and preoperative examination findings, operative times, postoperative hemogram values, postvoiding residual amounts and complications were examined.

In addition, FSI test results of women with sexual activity were compared with ICIQ-UI and UDI-6 interrogations related to urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* tlh operation with benign reasons and planned,
* concurrent stress describing urinary incontinence,
* Women between the ages of 40-65

Exclusion Criteria:

* planned operation with malignant causes,
* urinary tract infection,
* medication area for incontinence

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women between the ages of 40-65 who ; tlh operation with benign reasons and planned, and concurrent stress describing urinary incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
operation time | 2 years
  The duration of the procedure for stress urinary incontinence surgery was evaluated. recorded in minutes.
postoperative hemogram values | 2 years
  postoperative hemogram values were evaluated. Recorded in g / dl.
postvoiding residues | 2 years
  postvoiding residues were measured. Recorded in ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)